CLINICAL TRIAL: NCT03404154
Title: The Relation Between Endometrial Volume by 3D Vocal Ultrasound and Histopathology in Women With Postmenopausal Bleeding
Brief Title: Vocal in Assessment of Endometrium in Postmenopause
Status: Completed | Type: Observational
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other); om almasreen hospital ,Egypt (Unknown); National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: vocal
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Postmenopausal Bleeding
MeSH Terms: interventions — Dilatation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples Without DNA — Dilatation and curettage endometrial biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 3D ultrasound — it describes the diagnostic test which is 3D us to diagnose the cause of postmenopausal bleeding
Procedure: Dilatation and curretage — it describes the surgical maneuver that will be made to diagnose cause of bleeding

SUMMARY:
The unbalanced estrogen with no progesterone will lead to endometrial thickening .This thickening result in endometrial hyperplasia & carcinoma and lead to irregular bleeding

DETAILED DESCRIPTION:
Recent advances in the screening and diagnosis of endometrial pathologies (eg,endometrial hyperplasia , endometrial carcinoma ,endometrial polyps and myomas ) are directed towards non invasive methods as Transvaginal ultrasound with 3 D application using different softwares .

One of the applications of 3D Transvaginal Ultrasonography is Vocal technique ( Virtual Organ Computer aided Analysis ) that can measure volume especially in tissues with irregular borders And this technology is considered to be superior than the conventional 2 D ultrasound . .

ELIGIBILITY:
Inclusion Criteria:

-Postmenopausal women who were Complaining of Post-menopausal vaginal bleeding.

Exclusion Criteria:

* Women with hormone replacement therapy.
* Women showing intra-cavitary fluid collection at ultrasound examination
* Women with other gynecological lesions in the pelvis other than the uterus
* Previous diagnosis of endometrial pathology.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women with vaginal bleeding
Study Population: Postmenopausal women who were Complaining of Post-menopausal vaginal bleeding.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-25 (Actual)

PRIMARY OUTCOMES:
the number of participants who where diagnosed by 3D vocal to have endometrial carcinoma | within 4 weeks
  it describes how many women will be properly diagnosed with carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No